CLINICAL TRIAL: NCT06266975
Title: Chronic Kidney Disease Patient in Chronic Myloied Leukemia
Status: Not yet recruiting | Type: Observational
Sponsor: Sahar Mohammed Gad (Other)
Responsible Party: Sponsor-Investigator, Sahar Mohammed Gad, doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: CKD pts in CML
Record Dates: First submitted 2023-11-03; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Chronic Myeloid Leukemia in Remission
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Biobsy from kidney — using tyrosine kinase inhibitors particulary imatinib in ttt CML patients
  Other Names: drug , tyrosine kinase inhibitors particulary imatinib in ttt CML patients

SUMMARY:
To study the Prevalence ,Characteristics and outcome of CKD in patiants with chronic myeloid leukemia .

DETAILED DESCRIPTION:
* Chronic myeloid leukemia (CML) is a cancer of bone marrow that leads to an increased number of white blood cells. CML is more prevalent in the elderly and is characterized by weight loss, tiredness, shortness of breath, excessive sweating, bone pain, and frequent infections. [1] According to the American Cancer Society's estimates, CML represents 15% of all new leukemia cases.[2] The global burden of disease (GBD) study 2015 revealed that leukemia was under the top ten leading causes of death globally.[3] However, the latest GBD study found a decrease in the age-standardized incidence rate and the death rate from 1990-2017.[4] This dramatic improvement in the overall survival and health-related quality of life among CML patients was attributed to the impact of new therapeutic strategies. Tyrosine kinase inhibitors (TKIs), particularly imatinib, emerged as a potential therapeutic agent for the treatment of CML, reducing epidemiological burden (incidence rate), and improve quality of life.[5]
* The definition and classification of chronic kidney disease (CKD) have evolved over time, but current international guidelines define this condition as decreased kidney function shown by glomerular filtration rate (GFR) of less than 60 mL/min per 1•73 m2, or markers of kidney damage, or both, of at least 3 months duration, regardless of the underlying cause[6] Diagnosis is commonly made after chance findings from screening tests (urinary dipstick or blood tests), or when symptoms become severe. The best available indicator of overall kidney function is GFR, which is measured either via exogenous markers (eg, DTPA, iohexol), or estimated using equations. Presence of proteinuria is associated with increased risk of progression of CKD and death. Presence of proteinuria is associated with increased risk of progression of CKD and death.[7,8] Kidney biopsy samples can show definitive evidence of CKD, through common changes such as glomerular sclerosis, tubular atrophy, and interstitial fibrosis. Complications include anaemia due to reduced production of erythropoietin by the kidney; reduced red blood cell survival and iron deficiency; and mineral bone disease caused by disturbed vitamin D, calcium, and phosphate metabolism.[9

ELIGIBILITY:
Inclusion Criteria:1_ Chronic myloid leukemia patiants who diagonised by biopsy , 2_ CBC.

-

Exclusion : 1_pts known to have CKD before diagnosed of CML. 2- known Diabetic pts 3-imaging suggestive CKD etiology rather than CML effect eg.PKD,renal stones,chronic pyelonephritis

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all sexes , adult , not diabetic , not known CKD before diagnosed of CML
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Chronic Kidney Disease Patient in Chronic Myloied Leukemia | basline
  Using Non Invasive or invasive Methods and correlation between lab and radiological methods to find and a relation between CML and CKD and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Ramadan, Principal Investigator — Assist; Mohamed Ramadan, Study Director — Assiut University

REFERENCES:
- [Background] Webster AC, Nagler EV, Morton RL, Masson P. Chronic Kidney Disease. Lancet. 2017 Mar 25;389(10075):1238-1252. doi: 10.1016/S0140-6736(16)32064-5. Epub 2016 Nov 23. PMID 27887750
- [Background] Fathallah-Shaykh SA, Flynn JT, Pierce CB, Abraham AG, Blydt-Hansen TD, Massengill SF, Moxey-Mims MM, Warady BA, Furth SL, Wong CS. Progression of pediatric CKD of nonglomerular origin in the CKiD cohort. Clin J Am Soc Nephrol. 2015 Apr 7;10(4):571-7. doi: 10.2215/CJN.07480714. Epub 2015 Jan 29. PMID 25635034